CLINICAL TRIAL: NCT03681795
Title: Exploration of Glutamatergic System With PET Radiotracer in Gilles de la Tourette Patients: Pilot Study (GlutaTour)
Acronym: GlutaTour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/15/7836; 2017-000816-40 (EudraCT Number)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; the glutamatergic system; PET-scan; physiopathology
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: compare PET-evaluated glutamaergic system activity ([18F]-FNM) between patients with Gilles de la Tourette and healthy volunteers paired in sex, age and manual laterality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Experimental): patients with Gilles de la Tourette syndrome
  Interventions: Diagnostic Test: Experimental MRI exam and PET scan exam with radiotracer
- Control (Experimental): healthy control
  Interventions: Diagnostic Test: Experimental MRI exam and PET scan exam with radiotracer

INTERVENTIONS:
Diagnostic Test: Experimental MRI exam and PET scan exam with radiotracer — MRI exam and PET scan exam with radiotracer

SUMMARY:
Gilles de la Tourette syndrome is a neuropsychiatric disorder characterized by motor and vocal tics often associated with psychiatric comorbidities (obsessive compulsive disorder, anxiety and depressive syndrome, impulsivity). The pathophysiology of Gilles de la Tourette syndrome remains unclear.

DETAILED DESCRIPTION:
Gilles de la Tourette syndrome is a neuropsychiatric disorder characterized by motor and vocal tics often associated with psychiatric comorbidities (obsessive compulsive disorder, anxiety and depressive syndrome, impulsivity). The pathophysiology of Gilles de la Tourette syndrome remains unclear. It would involve an alteration of striatal-cortico-thalamic cortical circuits resulting in dopaminergic dysfunction. But glutamatergic hypothesis is also discussed from pharmacological, biochemical and genetic arguments. Exploration of glutamatergic system can be done in humans in vivo using a new radiotracer: the [18F] FNM (Fluoroethylnormemantine), a derivative of memantine. In the present study, aim of the study 1) to show the glutamatergic system "in vivo" in patients with Tourette's syndrome and 2) to perform correlations between various motor and behavioral symptoms and the pattern of brain fixation for this radiotracer. To do that, a pilot study will be conducted in 12 patients with Tourette's who will be evaluated in terms of motor (tics) and behavioral (OCD, anxiety, depression, impulsivity) symptoms. Each patient will have a PET-scan exam and a brain MRI exam. Data analysis will be carried out from two different approaches: first by region of interest, and secondly, without topographic a priori with the Statistical Parametric Mapping (SPM) software.

ELIGIBILITY:
Inclusion Criteria:

* Gilles de la Tourette syndrome according to the American Psychiatric association criteria (5 th ed, American Psychiatric association (APA), 2013)
* Aged 18 and over
* Patients treated with 2nd-generation neuroleptics for at least 3months
* Signed consent form

Exclusion Criteria:

* contraindications for MRI exam
* claustrophobia
* person under exclusive period for another study
* pregnant women
* patients under non-authorized treatment (1rst generation neuroleptics) or non-treated by neuroleptics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficients | Day 1
  Correlation coefficients is determined between the fixation of the PET tracer and the Total Tic score (TTS - from 0 to 50) which reflects the severity of tics in patients (under the Yale Global Tic Severity Scale - YGTSS)(Leckman and al, 1989).

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Day 1
  This scale represents the severity of tics in patients, it is a scale composed of three subscales:
  * Motor tic severity from 0 to 25,
  * Vocal Tic severity from 0 to 25,
  * Overall Impairment from 0 to 50, which reflects the functional impairment score (under Yale Global Tic Severity Scale - YGTSS). This score assesses the repercussions of the syndrome on self-esteem, and the social, professional and family.
  For each of the sub-scales, tics are rated according to their number, frequency, intensity, complexity, interference with activities of everyday life.
  The sum of Motor Tic severity and Vocal Tic severity form the Total Tic score (0 to 50)
Yale Brown Obsessive Compulsive Scale (Y-BOCS) - II | Day 1
  Yale Brown Obsessive Compulsive Scale consists of 19 questions aimed at evaluating the severity, the impact on daily, social, family and professional life activities of OCD, the anxieties generated by OCD Higher values represent a worse outcome
Hospital Anxiety Depression | Day 1
  Hospital Anxiety Depression (from 0 to 42) which is a self-questionnaire of 14 items:
  * 7 items refer to anxiety,
  * 7 items refer to depression. Each item is scored from 0 to 3 This scale explores anxiety and depressive symptoms. Total the anxiety and depression side: maximum 21 points for each.
  Between 8 and 10: doubtful anxiety or depressive state. Beyond 10: certain anxiety or depression.
Barrat Impulsivity Scale 11 | Day 1
  Barrat Impulsivity Scale 11 is self-assessment scale with 34 items. It provides an assessment of impulsivity according to motor impulsivity, cognitive impulsivity and planning difficulty. Each item is scored on 4, the total score therefore varies from 0 to 120

CONTACTS AND LOCATIONS:
Overall Officials: Christine BREFEL-COURBON, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Pierre-Paul Riquet - CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No